CLINICAL TRIAL: NCT02065726
Title: Whey Protein Supplementation in Malnourished Cancer Patients: a Randomized, Controlled Trial
Brief Title: Whey Protein Supplementation in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Norgine (Industry); Akern Srl (Industry)
Responsible Party: Principal Investigator, Emanuele Cereda, Physician, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20130018046
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2018-06

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Whey Proteins; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whey protein (Experimental): Nutritional counseling + 20 g (2 x 10 g) of whey proteins (Prother® - Spepharm Italy)
  Interventions: Dietary Supplement: Whey protein
- Nutritional counseling (Active Comparator): Nutritional counseling
  Interventions: Other: Nutritional counseling

INTERVENTIONS:
Dietary Supplement: Whey protein — Nutritional counseling consists in a personalized dietary prescription and regular (monthly) dietetic advise by a registered dietician + 20 g (2 x 10 g) of whey proteins
  Other Names: Prother® (Spepharm Italy)
  Arms: Whey protein
Other: Nutritional counseling — Nutritional counseling consists in a personalized dietary prescription and regular (monthly) dietetic advise by a registered dietician
  Arms: Nutritional counseling

SUMMARY:
Nutritional derangements are very common in cancer patients and negatively affect survival, morbidity and quality of life. Intervention trials have demonstrated that nutritional counseling can improve energy balance, nutritional status and quality of life in patients undergoing chemo-radiotherapy. Oxidative stress plays a role in the tumor-cytotoxic effect of cancer chemotherapy and radiotherapy but may also play a role therapy-related adverse events such as an impairment of nutritional status and quality of life. The nutritional properties of whey protein have recently raised attention. In view of the high content in cysteine these proteins can positively stimulate the synthesis of glutathione which, in turn, could contribute to the modulation of whole-body and cellular redox state. However, evidence on the role of this dietary intervention in cancer patients is limited.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients (lung, gastric, pancreatic, breast, colon, esophageal)
* Eastern Cooperative Oncology Group performance status ≤ 2
* Weight loss >= 10% in the last 6 months
* Chemotherapy
* Written informed consent

Exclusion Criteria:

* Age < 18 years
* Ongoing artificial nutrition (enteral or parenteral)
* Unavailability to planned measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2014-02-25 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Body composition | 3 months
  Change in phase angle assessed by bioelectrical impedance vectorial analysis (BIVA)

SECONDARY OUTCOMES:
Body composition | 1 month
  Change in phase angle assessed by bioelectrical impedance vectorial analysis (BIVA)
Body weight | 3 months
  Change in body weight during the study (at 1 month and 3 months)
Quality of life | 3 months
  Change in quality of life during the study (at 1 month and 3 months) as assessed by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire version 3.0 [EORTC QLQ-C30]
Handgrip strength | 3 months
  Change in handgrip strength during the study (at 1 month and 3 months)

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Cereda, MD, PhD, Principal Investigator — 1Nutrition and Dietetics Service, Fondazione IRCCS Policlinico San Matteo, Pavia, Italy; Riccardo Caccialanza, MD, Study Director — 1Nutrition and Dietetics Service, Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
Locations (1):
- Nutrition and Dietetics Service, Fondazione IRCCS Policlinico San Matteo, Pavia, Italy, Pavia, Pavia, Italy

REFERENCES:
- [Background] Langius JA, Zandbergen MC, Eerenstein SE, van Tulder MW, Leemans CR, Kramer MH, Weijs PJ. Effect of nutritional interventions on nutritional status, quality of life and mortality in patients with head and neck cancer receiving (chemo)radiotherapy: a systematic review. Clin Nutr. 2013 Oct;32(5):671-8. doi: 10.1016/j.clnu.2013.06.012. Epub 2013 Jun 26. PMID 23845384
- [Background] Baldwin C, Spiro A, Ahern R, Emery PW. Oral nutritional interventions in malnourished patients with cancer: a systematic review and meta-analysis. J Natl Cancer Inst. 2012 Mar 7;104(5):371-85. doi: 10.1093/jnci/djr556. Epub 2012 Feb 15. PMID 22345712
- [Background] Bounous G. Whey protein concentrate (WPC) and glutathione modulation in cancer treatment. Anticancer Res. 2000 Nov-Dec;20(6C):4785-92. PMID 11205219
- [Background] Tozer RG, Tai P, Falconer W, Ducruet T, Karabadjian A, Bounous G, Molson JH, Droge W. Cysteine-rich protein reverses weight loss in lung cancer patients receiving chemotherapy or radiotherapy. Antioxid Redox Signal. 2008 Feb;10(2):395-402. doi: 10.1089/ars.2007.1919. PMID 18158761
- [Derived] Cereda E, Turri A, Klersy C, Cappello S, Ferrari A, Filippi AR, Brugnatelli S, Caraccia M, Chiellino S, Borioli V, Monaco T, Stella GM, Arcaini L, Benazzo M, Grugnetti G, Pedrazzoli P, Caccialanza R. Whey protein isolate supplementation improves body composition, muscle strength, and treatment tolerance in malnourished advanced cancer patients undergoing chemotherapy. Cancer Med. 2019 Nov;8(16):6923-6932. doi: 10.1002/cam4.2517. Epub 2019 Sep 30. PMID 31568698